CLINICAL TRIAL: NCT03511963
Title: A Randomized, Double-blind, Parallel Control, Multicenter, Phase III Clinical Study to Compare the Efficacy and to Evaluate the Safety and Immunogenicity of HLX04 and Bevacizumab Combined With Oxaliplatin and Fluoropyrimidine-based Chemotherapy (XELOX or mFOLFOX6) in the First-line Treatment of Metastatic Colorectal Cancer (mCRC)
Brief Title: A Clinical Study to Compare the Efficacy, Safety and Immunogenicity of HLX04 and Bevacizumab Combined XELOX or mFOLFOX6 in the First-line Treatment of mCRC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX04 mCRC03
Record Dates: First submitted 2018-03-21; First posted 2018-04-30 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Injections; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX04 (Experimental)
  Interventions: Drug: HLX04 100 mg in 4 ml Injection
- Bevacizumab (Active Comparator)
  Interventions: Drug: Avastin 100 mg in 4 ml Injection

INTERVENTIONS:
Drug: HLX04 100 mg in 4 ml Injection — 7.5 mg/kg iv (XELOX+HLX04) 5 mg/kg iv (mFOLFOX6 + HLX04)
  Arms: HLX04
Drug: Avastin 100 mg in 4 ml Injection — 7.5 mg/kg iv (XELOX+HLX04) 5 mg/kg iv (mFOLFOX6 + HLX04)
  Arms: Bevacizumab

SUMMARY:
This trial is conducted in patients with the recurrent lesion(s) post-surgery or the untreated mCRC. After stratification with respect to ECOG PS score, chemo regimen, primary tumor location and KRAS and BRAF genotype (complete wild-type/primal type), eligible patients are randomized into two arms at 1:1 ratio to receive HLX04 (Arm A) or Bevacizumab (Arm B) in combination with one of the protocol-defined chemotherapies, modified FOLFOX6 (mFOLFOX6) or XELOX for mCRC until disease progression (PD) or unacceptable toxicity or achieving an operable contingency, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
3. Life expectancy ≥ 6 months
4. Histologically confirmed colorectal cancer with a metastatic / recurrent lesion that cannot be cured by surgery.
5. At least one measurable lesion have been the confirmatory detection within 4 weeks prior to the randomization with respect to RECIST 1.1
6. No prior first-line systemic anti-tumor therapy for mCRC (including systemic chemotherapy, molecular targeted therapy, biotherapy, and other study treatment) have been identified
7. At least 6 months have elapsed if considering the interval from the time of firstly documented metastasis to the post-operational adjuvant chemotherapy termination
8. Adequate organ function as indicated by the following laboratory values:

   1. Absolute neutrophil count (ANC) ≥1,500 /mm3（1.5×109 /L）
   2. Platelets ≥80,000 / mm3（80×109 /L）
   3. Hemoglobin ≥9 g/dL, within the 2 weeks prior to the screening no need for the transfusion
   4. Serum creatinine ≤1.5 X upper limit of the normal (ULN) or creatinine clearance ≥ 50 mL/min according to Cockcroft-Gault formula
   5. Serum total bilirubin ≤ 1.5 X ULN
   6. AST (SGOT), ALT (SGPT) and alkaline phosphatase (ALK) ≤ 3 X ULN (AST/ALT ≤ 5 X ULN if liver metastatic; ALK ≤ 5 × ULN if liver and/or bone metastastic)
   7. International Normalized Ratio (INR) or Prothrombin Time (PT) or Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN; ( if patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intent using goal of anticoagulants)
9. The subjects are accredited with good compliance, signed the informed consent, and capable to cooperate, completing the relevant examination and follow-ups.

Exclusion Criteria:

1. Targeted medicine(including Bevacizumab, cetuximab, panedol, arbicip, rigofeni, etc) was used before as adjuvant therapy.
2. Cerebral and/or leptomeningeal metastasis.
3. Bleeding predisposition, high bleeding risk or coagulant disorder, thrombotic event(s) occurrence ≤6 months and/or hemoptysis ≤3 months (≥ 1/2 teaspoons fresh blood each) prior to the screening; use of full dose oral or parenteral anticoagulant or thrombolytic medication (allowing preventative anticoagulation); use of aspirin (> 325 mg/day) or other platelet-inhibition non-steroidal anti-inflammatory drugs within 10 days since the screening; CT/MRI imaging evidence, testimony of the main arteries/veins (such as pulmonary artery or superior vena cava) being infringed, encroached.
4. Subjects with uncontrolled hypertension and with a medical history of hypertensive crisis or hypertensive encephalopathy; serious cardiovascular and cerebrovascular diseases, including cerebrovascular accident (CVA) ≤6 months before the screening, transient ischemic attack (TIA), myocardial infarction and significant vascular disease (including but not limited to aortic aneurysms with need for surgical repair or recent evidence of arterial thrombosis), unstable angina, heart failure and serious arrhythmias that are uncontrolled by drugs (New York Heart Association Class ≥2).
5. Subjects with non-healing wounds, active peptic ulcer or fracture and active infection; tracheal esophageal fistula, gastrointestinal perforation or gastrointestinal fistula and abdominal abscess in the 6 months prior to the screening;Uncontrolled infection,including HIV,HBV,HCV and syphilis .
6. Subjects allergic to bevacizumab, oxaliplatin, 5-FU/capecitabine or folinic acid injection and the relevant ingredients and excipients.
7. Pregnant women and lactating women; women of potential childbearing age and male subjects do not use effective contraception during the study period, and during the 6 months after the last study drug administration effective contraception cannot be assured.
8. Presence of other active malignancies or a history of other malignancies within the past 5 years, except for carcinoma in situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin that has been previously treated with curative intent.
9. Subject is currently enrolled in, or ≤4 weeks since subject participating another investigational device or drug study(s), or subject is receiving other investigational agent(s).
10. Any other medical condition that renders disqualification for the inclusion in the study according to the investigator discretionary judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
PFSR9m | 0 to 36 weeks
  Progression free survival rate (PFS rate) at Month 9 (PFSR9m)

SECONDARY OUTCOMES:
BORR | 0 to 48 weeks
  Best objective response rate (BORR) up to Week 48
ORR | 6 to 48 weeks
  Objective response rate (ORR) at Weeks 6, 12, 18, 24, 36，42,48
OSR | 0 to 48 weeks
  Overal survival rate: the time from the date of randomization to the date of documented clinical or radiological progression or death due to any cause within 48 weeks after first visit
TTR | 0-48 weeks
  Time to response (TTR)
DOR | 0-48 weeks
  Duration of response (DOR)
SAE | 0-48 weeks
  incidence of serious adverse events (SAE)

OTHER OUTCOMES:
Cmax | 0 to 54 weeks
  Cmax following first dose and the dose of Week 18;
Ctrough | 0 to 54 weeks
  Ctrough before the first dose of Cycle2, Week 18, Week 36;

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Bayi Hospital Ethics Committee, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhu X, Qian H, Sun J, Wu M, Yu C, Ding Y, Zhang X, Chai K, Li X. A phase 1 randomized study compare the pharmacokinetics, safety and immunogenicity of HLX04 to reference bevacizumab sourced from the United States, the European Union, and China in healthy Chinese male volunteers. Cancer Chemother Pharmacol. 2021 Sep;88(3):465-474. doi: 10.1007/s00280-021-04297-z. Epub 2021 Jun 4. PMID 34086067
- [Derived] Qin S, Li J, Bai Y, Shu Y, Li W, Yin X, Cheng Y, Sun G, Deng Y, Zhong H, Li Y, Qian X, Zhang L, Zhang J, Chen K, Kang W; HLX04-mCRC03 Investigators. Efficacy, Safety, and Immunogenicity of HLX04 Versus Reference Bevacizumab in Combination with XELOX or mFOLFOX6 as First-Line Treatment for Metastatic Colorectal Cancer: Results of a Randomized, Double-Blind Phase III Study. BioDrugs. 2021 Jul;35(4):445-458. doi: 10.1007/s40259-021-00484-9. Epub 2021 May 20. PMID 34014555
- See also: Related Info — http://doi.org/10.1016/j.annonc.2020.10.124